CLINICAL TRIAL: NCT03051737
Title: Development and Validation of a Regional Multi-scale System in Ile-de-France for the Prediction of the Patient Flow in the Emergency Department and the Need for Hospitalization
Brief Title: Development and Validation of a Regional Multi-scale System for the Prediction of the Patient Flow in the Emergencies and the Need for Hospitalization
Acronym: PRED-URG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI15018
Record Dates: First submitted 2017-02-06; First posted 2017-02-14 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Emergency Department; Hospitalization
Keywords: Multi-scale; Prediction; Patient Flow; Emergency Department; Hospitalization; Ile-de-France
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this retrospective study is to validate a prediction system of emergencies department (ED) attendance on a wide range of time and the need for hospitalization, at various levels of perimeter (with all emergency departments or one ED in particular), with all patients or with one sub-group of patients (age, gravity, care).

DETAILED DESCRIPTION:
As secondary objectives, the study aims:

* to measure the influence of different factors as environmental or structural and to identify the modifiable factors, then to allow us to test by simulation, impact of various interventions (for example: opening of hospitals and reinforcement of ED teams) on arrival flows or regenerated tension inside ED teams.
* to study the relation between the flows (arrival patients, hospitalized patients) and the time of ED visit or the indicators of tension of ED team.
* Typology of ED in the region of Paris permitting afterward comparison the benchmarking type between similar structures.

This retrospective study will be performed on database: individual data in the region of Paris of summation of ED visits and data on the structures of health cares, as well as environmental data (principal given cares, weather, moves, circulations, pollution, strikes, vacations, etc.)

ELIGIBILITY:
Inclusion Criteria:

* All subjects have been recorded as patients in emergency departments between 2010 and 2015.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults or children who have been recorded as patients in emergency departments between 2010 and 2015 are all eligibles with unlimited number of care.
  85 Health Facilities in Ile de France who have emergency departments will participate the study.
Sampling Method: Non-Probability Sample
Enrollment: 18000000 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Prediction of emergency department visits | throughout the study, an average of 18 months
  Calculated base on regional database: individual data of summation of ED visits in the region of Paris and structural data of health cares

SECONDARY OUTCOMES:
Prediction by age | throughout the study, an average of 18 months
  By sub-group of child or senior
Prediction by lever of gravity | throughout the study, an average of 18 months
Prediction by type of care | throughout the study, an average of 18 months
  By type : (medical, surgical or intensive) care
Prediction by need of hospitalization or no | throughout the study, an average of 18 months
Relation between flow of patients and indicator of tension of team | throughout the study, an average of 18 months
Relation between flow of patients and time of ED visit | throughout the study, an average of 18 months
Typology of ED of the region of Paris | throughout the study, an average of 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Mathias WARGON, MD, Principal Investigator — Emergency Department - Bry sur Marne Hospital
Locations (1):
- Emergency Department - Bry sur Marne Hospital, Bry-sur-Marne, Val-de-Marne, France

IPD SHARING:
Plan to Share IPD: No